CLINICAL TRIAL: NCT05278806
Title: Evaluating the Impact of an Equity Focused Dashboard and Clinical Support on Disparities in Primary Care Ambulatory Quality Outcome Measures: a Quality Improvement Research Project
Brief Title: Evaluating the Impact of an Equity Focused Dashboard and Clinical Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew S. Hwang, M.D., Assistant Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P000354
Record Dates: First submitted 2021-11-09; First posted 2022-03-14 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Hypertension; Diabetes; Breast Cancer
Keywords: Equity; Health Disparities
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Equity Dashboard, Population Health Coordinator and Community Health Worker Support (Experimental): After the step in which the primary care providers are randomized to receiving intervention, one group of providers will receive the equity dashboard data and complete an equity huddle where they will review their list of eligible patients (Black, Indigenous and People of Color [BIPOC] patients and patients with limited English proficiency [LEP]) with a population health coordinator (PHC). The goal of the equity huddle will be to develop a plan to improve eligible patients' hypertension control. One of the options will be to refer patients to a community health worker (CHW) program focused specifically on addressing hypertension.
  Interventions: Other: Equity Dashboard, Population Health Coordinator and Community Health Worker Support
- Equity Dashboard and Population Health Coordinator Support (Experimental): After the step in which the primary care providers are randomized to receiving intervention, a second group of providers will receive the equity dashboard data and complete an equity huddle where they will review their list of eligible patients (Black, Indigenous and People of Color [BIPOC] patients and patients with limited English proficiency [LEP]) with a population health coordinator (PHC). The goal of the equity huddle will be to develop a plan to improve eligible patients' hypertension control.
  Interventions: Other: Equity Dashboard and Population Health Coordinator Support
- Delayed intervention (No Intervention): Black, Indigenous and People of Color (BIPOC) patients and patients with limited English proficiency (LEP) before their primary care providers are randomized to receiving the intervention. (By the end of the 12 steps, all BIPOC/LEP patients will be assigned to an experimental group)
- Usual Care (No Intervention): Patients who are not eligible for additional clinical support (i.e. White and English speaking patients).

INTERVENTIONS:
Other: Equity Dashboard, Population Health Coordinator and Community Health Worker Support — Providers will be given access to an equity dashboard that displays their practice's performance on ambulatory quality metrics stratified by race and language.
  Population health coordinators (PHCs) will lead equity huddles with providers to review list of patients who are not at goal for their hypertension control and meet the inclusion criteria. Providers will formulate a follow up plan for each patient that the PHCs will help implement. For example, PHCs may contact patient via the online patient portal or phone to obtain recent home blood pressure readings, facilitate scheduling of follow up visits, etc.
  In addition, patients may be referred to the community health worker (CHW) hypertension management program. Patients will work with the CHW for 3-6 months. During this time the CHW will focus their efforts on patient education/coaching, remote blood pressure monitoring, addressing psychosocial and socioeconomic barriers to care and care coordination.
  Arms: Equity Dashboard, Population Health Coordinator and Community Health Worker Support
Other: Equity Dashboard and Population Health Coordinator Support — Providers will be given access to an equity dashboard that displays their practice's performance on ambulatory quality metrics stratified by race and language.
  In addition, population health coordinators (PHCs) will lead disparities focused huddles with providers. During the huddle, they will review list of patients who are not at goal for their hypertension control and meet the inclusion criteria. Providers will then formulate a follow up plan for each patient that the Population Health Coordinators will help implement. For example, PHCs may contact patient via the online patient portal or phone to obtain recent home blood pressure readings, facilitate scheduling of follow up visits, etc.
  Arms: Equity Dashboard and Population Health Coordinator Support

SUMMARY:
In this project, the impact of providing a practice-level equity dashboard that displays ambulatory quality outcome metrics stratified by race and language to primary care providers at Massachusetts General Hospital (MGH) will be evaluated. Provision of the dashboard data will be paired with additional clinical support focused on hypertension control among Black, Indigenous and People of Color (BIPOC) and patients with limited English proficiency (LEP).

The investigators hypothesize that there will be a improvement in hypertension control (primary outcome), diabetes control and breast cancer screening (secondary outcomes) among Black, Indigenous and People of Color (BIPOC) and patients with limited English proficiency (LEP) in the intervention period compared to the control period.

DETAILED DESCRIPTION:
A clinical program will be implemented to utilize the equity dashboard in routine clinical practice augmented by clinical support to address current disparities in hypertension control among MGH primary care patients who are Black, Indigenous and People of Color (BIPOC) as well as patients with limited English proficiency (LEP). The clinical support will be provided by population health coordinators (PHCs) and/or community health workers (CHWs).

To evaluate the program, the investigators propose a stepped wedge design that will randomize the primary care providers to the provision of the equity dashboard and additional clinical support at different intervals. The primary reason to randomize the primary care providers is because the PHCs and CHWs have limited capacity to contact and assist the patients in our primary care practices with poorly controlled hypertension and can only engage a limited number of patients at a time.

The stepped wedge cluster-randomized study design will randomize providers in all 15 MGH primary care practices to receiving the intervention (i.e. equity dashboard with additional clinical support) in twelve groups. Each step will be a one-month period. Providers randomized to Group 1 will receive the equity dashboard data as well as additional clinical support starting in Step 1 while providers randomized to Group 12 will receive the same intervention at the beginning of Step 12 but receive usual care in Steps 0-11. We will match Providers in the opposite steps (e.g. Group 1 vs. Group 12, Group 2 vs. Group 11, etc.) by practice, baseline hypertension control rate, and the number of patients in their panel who are eligible for the intervention to ensure balance between data collected from the intervention periods and control periods. The stepped wedge design will allow for an open cohort (i.e. new patients of the providers allocated to the intervention can enter in subsequent steps) and a repeated measures data analysis with the same patients experiencing both control and intervention conditions.

ELIGIBILITY:
<Provider Eligibility>

Inclusion Criteria:

• Massachusetts General Hospital primary care physician

Exclusion Criteria:

• Practice leaders and equity steering committee members as they will all get access to the equity dashboard data.

<Patient Eligibility>

Inclusion Criteria:

• Uncontrolled Hypertension AND Black, Indigenous and People of Color (BIPOC) patients or Limited English proficiency (LEP).

Exclusion Criteria:

• Not deemed appropriate for intervention by their primary care provider due to terminal illness, advanced dementia, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10766 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Hypertension control | 1 year
  * Blood pressure (BP) measured in the last 12 months AND last BP or average of last three BP readings (in the last 18 months) <130/80 or
  * BP measured within past 6 months AND either the last or average of last three BP readings (in the last 18 months) meet one of the following criteria:
    * Age < 60, BP ≤ 140/90
    * Age ≥ 60 with Diabetes, BP ≤ 140/90; without Diabetes, BP ≤ 150/90
    * Age ≥ 60, Diastolic BP < 70, regardless of Systolic
    * On three or more anti-hypertensive medications from three different classes

SECONDARY OUTCOMES:
Hemoglobin A1c control | 1 year
  * Most recent HbA1C in the last 12 months was <7.0% OR
  * Most recent HbA1C within the last 6 months was ≤ 9.0%
Breast cancer screening rates | 1 year
  Completed a mammogram in the past 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Hwang, MD/MPH, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang AS, Chang Y, Matathia S, Brodney S, Barry MJ, Horn DM. Effectiveness of a Population Health Intervention on Disparities in Hypertension Control: A Stepped Wedge Cluster Randomized Clinical Trial. J Gen Intern Med. 2024 Nov;39(15):3028-3034. doi: 10.1007/s11606-024-08839-y. Epub 2024 Jun 12. PMID 38865006